CLINICAL TRIAL: NCT01345617
Title: A Study of Sweat Testing Using a Quantitative Patch
Status: Completed | Type: Observational
Sponsor: Polychrome Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011-0291; CFQuantum001 (Other: PolyChrome Medical, Inc.)
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cystic fibrosis patients: cystic fibrosis patients
- non-cystic fibrosis patients: non-cystic fibrosis patients

SUMMARY:
The primary aim of the study is to determine if the CF Quantum Sweat Test provides sweat chloride results that are equivalent to the results from traditional sweat testing. The secondary aim of the study is to assess the quantity not sufficient rate of the CF Quantum Sweat Test compared to traditional sweat testing.

DETAILED DESCRIPTION:
All 50 states and the District of Columbia are performing newborn screening for cystic fibrosis (CF). Infants who have a positive newborn screen require follow-up with a sweat test. Gibson-Cooke Quantitative Pilocarpine Iontophoresis (GCQPIT) requires collecting sweat in microbore tubing or on gauze/filter paper and analyzing sweat using a chloridometer. This test has many difficulties including specimens that are quantity not sufficient (QNS), many steps of pipetting solutions in the laboratory, and the need for a chloridometer to analyze sweat chloride concentration. The only manufacturer of a chloridometer has ceased production of this instrument. The CF Quantum® Sweat Test System (CFQT) overcomes all of the difficulties of GCQPIT. This pilot study will determine if the CFQT provides results that are equivalent to GCQPIT.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cystic fibrosis
* patients who require a sweat test

Exclusion Criteria:

* Infants less than 48 hours of age
* Patient is receiving oxygen by open delivery
* collection site has diffuse inflammation or rash

Min Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pediatric pulmonology clinic
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
sweat chloride value | once, at enrollment (baseline)
  Sweat chloride measurements obtained by GCQPIT and CFQT

SECONDARY OUTCOMES:
QNS rate | once, at enrollment (baseline)
  QNS rate of CFQT compared to GCQPIT

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Rock, MD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - University of Utah, Salt Lake City, Utah
  - American Family Children's Hospital, Madison, Wisconsin